CLINICAL TRIAL: NCT05360745
Title: Study of the Impact on Quality of Life of Nutritional Supplementation With a Food Supplement Versus Placebo in Patients With Locally Advanced/Metastatic Pancreatic Cancer.
Brief Title: Quality of Life With Nutritional Supplementation in Patients With Locally Advanced/Metastatic Pancreatic Cancer.
Acronym: FOODPANC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Few months later the site initiation visit, the principal investigator decided not to continue with the study. He explained that his investigational team was not able to combine the study procedures with their usual clinical practice.
Sponsor: Fundacion para la Excelencia y la Calidad de la Oncologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: fe-2021-001
Record Dates: First submitted 2022-04-20; First posted 2022-05-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Quality of Life; Locally Advanced Pancreatic Carcinoma; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): ARACOMPLEX® (food supplement). 2 tablets per day, during 6 months.
  Interventions: Dietary Supplement: ARACOMPLEX®
- Control arm (Placebo Comparator): Placebo. 2 tablets per day, during 6 months.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: ARACOMPLEX® — ARACOMPLEX® is an authorized food supplement that contains maca extract, vitamin complexes and ions, and that improves the quality of life of the patient.
  Arms: Experimental arm
Dietary Supplement: placebo — Placebo has a composition that makes its weight and organoleptic characteristics are identical to ARACOMPLEX®.
  Arms: Control arm

SUMMARY:
Metastatic pancreatic cancer has a poor prognosis, with approximately one-third of patients experiencing poor quality of life at six months.

ARACOMPLEX® is a food supplement that contains maca extract, vitamin complexes and ions, and this nutritional contribution seems to favor the improvement of the patient's quality of life. To verify this statement, this experimental study is carried out in patients with locally advanced/metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This study is composed of two phases: pilot phase and experimental phase. The pilot phase is also composed of two stages: first stage of pilot phase and second stage of pilot phase.

There are 22 patients recruited within the first stage of the pilot phase. 11 patients will be treated with ARACOMPLEX® and 11 patients will be treated with placebo. If the results are positive, a second stage of the pilot phase will take place until 43 patients are recruited in each treatment group, that is, 32 more patients in each group. The placebo group in the pilot phase is not analyzed.

In the experimental phase, a total of 234 patients are required, that is, 117 patients in each of the two study groups (ARACOMPLEX® and placebo). This phase will include the patients who participated in the pilot phase (86 patients, 43 randomized patients in each group) and 148 additional patients (74 patients in each group) up to a total of 234 patients (117 patients in each group).

If the results obtained from the analysis of the data from the first stage of the pilot phase are satisfactory, according to the protocol, the sponsor will present these results to the ethics committee, at the same time that also an addition of investigational sites, to move on to the second stage of the pilot phase. The approval or authorization of the ethics committee is required to progress to the second stage of the pilot phase.

The criteria for moving to the second stage is that more than 7 responders patients are achieved, after 6 months of treatment, out of the 11 patients in the experimental group. The responder patient is the one who meets an improvement in quality of life (difference of at least 10 points of quality improvement on the EORTC QLQ-C30 scale) between baseline and final time.

If the expected successful results are not obtained, the study will be closed and a new study will be proposed based on the data provided at this stage.

If the results obtained from the data analysis from the second stage of the pilot phase are satisfactory, according to the protocol, the sponsor will present these results to the ethics committee, at the same time as also an addition of investigational sites, if applicable. The ethics committee will be responsible for authorizing or approving the transition from the second stage of the pilot phase to the experimental phase.

The criteria for moving on to the experimental phase is that more than 30 responders patients are achieved, after 6 months of treatment, out of the 43 patients in the experimental group. The responder patient is the one who meets an improvement in quality of life (difference of at least 10 points of quality improvement on the EORTC QLQ-C30 scale) between baseline and final time.

In this study, the data of the patients included in the pilot phase will be counted, that is, the data of the 86 patients (ARACOMPLEX® and placebo), for which 148 additional patients are required in this phase (74 more patients in the ARACOMPLEX® group and 74 more in the placebo group) to reach a total of 234 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with locally advanced or metastatic pancreatic cancer without previous chemotherapy treatment.
* Patients for whom chemotherapy treatment has been indicated.
* Adequate bone marrow function (neutrophils ≥1500 mm3, platelets ≥100,000 mm3), adequate liver function (bilirubin ≤1.5 times the upper limit of the normal range)
* Adequate renal function (glomerular filtration rate greater than or equal to 90 ml/min/1.73).
* ECOG functional stage 0-1 (Karnofsky ≥ 80).
* Patients must agree to carry out study visits and procedures with precise instructions.

Exclusion Criteria:.

* Age ≥76 years.
* Endocrine or acinar pancreatic cancer.
* Serious systemic diseases such as: sepsis, heart failure, severe COPD, liver failure and chronic kidney disease.
* Prior radiation to areas of measurable disease.
* Chronic diarrhea.
* Active infection.
* Significant medical history of heart disease.
* Pregnancy or lactation.
* Impossibility of the patient, due to medical condition, to follow the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | 6 months
  To assess the degradation of quality of life at 6 months using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale in patients with locally advanced/metastatic pancreatic cancer receiving chemotherapy and supplementation with ARACOMPLEX® (PILOT PHASE) and compared with patients that are treated with chemotherapy and placebo (EXPERIMENTAL PHASE).
  The EORTC QLQ-C30 includes the "Global Health Status/Quality of life" scales, which are composed by items 29 and 30, and they are scored from 0 (worse) to 100 (better).

SECONDARY OUTCOMES:
Nutritional status assessment | Baseline, 1 month, 3 months and 6 months.
  Measured by the Malnutrition Screening Tool (MST)
Functional status assessment | Baseline, 1 month, 3 months and 6 months.
  Measured by the Eastern Cooperative Oncology Group (ECOG) scale. The score is from 0 (better) to 5 (worse outcome, death)
Functional status assessment | Baseline, 1 month, 3 months and 6 months.
  Measured by the Karnofsky scale.The score is from 100 %, normal activity and no evidence of disease, to 0 %, dead. Values ≤ 40% mean that patient is unable to care for self and requires equivalent of institutional or hospital care; diseases may be progressing rapidly.
Tumor response assessment | Assessment at the end of the third and sixth chemotherapy cycles, as per normal clinical practice.
  Measured by the RECIST criteria v.1.1
Compliance treatment | 1 month, 3 months and 6 months.
  Measured as the percentage of tablets taken from the previous visit: (number of tablets taken since the last visit (n) / number of days since the last visit (N) ) x 100.
Adverse events due to chemotherapy | 1 month, 3 months and 6 months.
  The assessment of adverse events due to chemotherapy is performed according to the CTCAE criteria, and are those reported as per usual clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Sandiego, Doctor, Principal Investigator — Fundación Instituto Valenciano de Oncología

IPD SHARING:
Plan to Share IPD: No